CLINICAL TRIAL: NCT06854341
Title: A Canadian Retrospective Analysis of Persistence on Ofatumumab Using Patient Support Program Data
Brief Title: A Canadian Study of Persistence on Ofatumumab Using Patient Support Program Data
Acronym: CAPES
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GCA04
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Patient Support Program; Ofatumumab; Persistence
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Ofatumumab Cohort: Adult patients with relapsing remitting multiple sclerosis (RRMS) who started treatment with ofatumumab, and were enrolled in the Kesimpta Go Program.

SUMMARY:
This was an observational, non-interventional, real world study involving secondary use of de-identified aggregate data from patients prescribed ofatumumab, collected by the Kesimpta Go Program in Canada. This study utilized a cohort design. The study period included all available data captured by the Kesimpta Go Program from program inception (April 2, 2021) to the time of data transfer (May 1, 2024). Patients were indexed into the study on the date they started their medication, from April 2, 2021 to May 1, 2024. The baseline period represented the period prior to ofatumumab treatment initiation. Baseline variables were collected from the enrollment form, which include demographic and clinical history, such as whether the patient had prior treatment with disease-modifying therapy (DMT). Patients were followed until the first of the following censoring events: ofatumumab discontinuation; end of the study period; or leaving the Kesimpta Go Program.

ELIGIBILITY:
Inclusion criteria:

Patients were included if they met all of the following criteria:

* Patients enrolled in the Kesimpta Go Program
* Patients with documented informed consent from enrollment in the Kesimpta Go Program
* Patients who started treatment with ofatumumab

Exclusion criteria:

Patients were excluded if they met any of the criteria below:

* Patients with no demographic information
* Patients who could not be linked across the data sources required for analysis (Kesimpta Go Program Enrollment Form, Pharmacy Claims Forms, Kesimpta Go Program Database)
* Patients with 3+ treatment interruptions (patient was "on hold" - i.e., not currently receiving the treatment in the patient support program)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, non-interventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 5448 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients who Discontinued Ofatumumab per Patient Characteristic | Month 6, 12, 18, 24, 30, and 36
  Patient characteristics included age group, gender, type of insurance, and experience (naive or experienced) of disease-modifying therapy (DMT) before starting ofatumumab.

SECONDARY OUTCOMES:
Number of Patients per Demographic Category | Baseline
  Demographic categories included age, age group, gender, index year, and type of insurance. Index year was the year patients started their medication.
Number of Patients per Clinical History Characteristic | Baseline
  Clinical history characteristics included experience of disease-modifying therapy (DMT) before starting ofatumumab (naive or experienced) and the type of last DMT used before starting ofatumumab.
Cox Proportional Hazard Ratio for the Association Between Discontinuation of Ofatumumab and Patient Characteristics | Up to 3 years
  Patient characteristics included age group, gender, type of insurance, and type of last DMT used before starting ofatumumab.
Number of Patients by Reason for Discontinuation of Ofatumumab Treatment | Up to 3 years
  Reasons for discontinuation included lack of efficacy, non-adherence, side effects, switched medications, trying to conceive/pregnancy, patient request, physician request, treatment interruption gap >90 days.
Number of Patients by Reason for Leaving the Kesimpta Go Program | Up to 3 years
  Reasons for leaving the Kesimpta Go program included could not contact participant, deceased, doesn't meet eligibility, patient moved, refused coverage, reimbursement issues, no reason given.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Selchen D, Grant R, Magnussen C, Murray J, Neish CS. A real-world study on persistence with ofatumumab in Canadian patients with multiple sclerosis. Mult Scler Relat Disord. 2026 Jan 6;107:106976. doi: 10.1016/j.msard.2026.106976. Online ahead of print. PMID 41529661
- See also: Results for COMB157GCA04 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18277